CLINICAL TRIAL: NCT02540044
Title: Supporting Patient Care With Electronic Resource (SuPER): Efficacy of an Online Decision Aid for Patients Considering Biologic Therapy for Rheumatoid Arthritis
Brief Title: Supporting Patient Care With Electronic Resource (SuPER)
Acronym: SuPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Alberta (Other); Simon Fraser University (Other); Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H15-02046
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANSWER-2 decision aid (Experimental): The Intervention Group will receive simple instructions to access ANSWER-2 and complete the program on their own computers within two days. At the end of the session, ANSWER-2 will produce a one-page summary summarizing the participant's questions, concerns, and preferred medication option.
  Interventions: Behavioral: ANSWER-2 decision aid
- Control Group (TAS Consumer Guide) (Active Comparator): The Control Group will receive the online Arthritis Medications: A Consumer's Guide, published by The Arthritis Society. It contains standard information about biologics, including an introduction of the different biologic options, dosages and side effects.
  Interventions: Behavioral: Control Group (TAS Consumer Guide)

INTERVENTIONS:
Behavioral: ANSWER-2 decision aid — ANSWER-2 will consist of: 1) an Information Module that presents effectiveness and side effects of each treatment option, and 2) an interactive Value Clarification Module that guides patients to consider what matter to them the most, and the pros and cons of each treatment option. Within the Information Module, the decision support information (i.e., the benefits and harms of treatment options) will be presented in narrated text, graphics, and a series of animated patient stories demonstrating attributes required for effective communication with doctors and significant others.
  Arms: ANSWER-2 decision aid
Behavioral: Control Group (TAS Consumer Guide) — The Arthritis Society Consumer guide pdf.
  Arms: Control Group (TAS Consumer Guide)

SUMMARY:
This proof-of-concept randomized trial evaluates the effectiveness of using an on-line decision aid (ANSWER-2) in the decision making to start or switch biologic therapy in Canadian patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The proposed project aims to improve the process of making evidence-informed treatment decisions by patients with rheumatoid arthritis (RA) and ultimately, empower patient self-management. Current RA treatment emphasizes: 1) the need for early and aggressive treatment, and 2) the use of a Treat-to-Target approach. Patients often struggle with treatment decisions, however, especially when the options have both benefits and risks. To address this challenge, the investigators have developed a new online decision aid called ANSWER-2 (ANimated, Self-serve, WEb-based, Research Tool: Version 2) for RA patients who are considering a biologic or other new therapy. A unique feature of ANSWER-2 is its ability to individualize how treatment options are presented based on the patient's preferences.

Objective: 1) To evaluate the effectiveness of ANSWER-2 in reducing patients' decisional conflict. 2) To assess the extent to which ANSWER-2 improves patients' knowledge about RA medications and confidence in managing their health. 3) To examine the experiences of patients and rheumatologists in using the ANSWER-2.

The investigators will conduct a proof-of-concept randomized controlled trial with 148 patients with RA. Eligible individuals are those: 1) with a diagnosis of RA from a rheumatologist, 2) whose rheumatologists have recommended initiating a biologic or other new therapy or switching to another agent, and 3) who have internet access. The Intervention Group will receive simple instructions to access ANSWER-2 and complete the program on their own within two days. At the end of the session, a one-page summary will be produced to help them discuss their questions, concerns, and preferred choices with their health care providers. The Control Group will receive The Arthritis Society's online education booklet "Arthritis Medications: A Consumer's Guide". Participants will complete the Decisional Conflict Scale (primary outcome) before and after the intervention (ANSWER-2 or booklet). The following secondary outcome measures will be collected at baseline, 1 month and 2 months: 1) Medication Education Impact Questionnaire (MeIQ), and 2) Partners in Health Scale (PHS). In addition, use of healthcare resources will be collected at 2 months. Participants will also be asked about their medication preferences at Month 1, as well as the shared decision making process in their last appointment, (using the 3-item CollaboRATE scale), at Month 1. Participants who received the ANSWER-2 decision aid and their rheumatologists will be invited to participate in an interview about their experience with the patient decision aid. The investigators will use analysis of variance (ANOVA) to compare between the Intervention Group and Control Group, using the baseline measure as a covariate. An iterative content analysis will be conducted for the qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are as follows: 1) with a diagnosis of RA from a rheumatologist, 2) whose rheumatologists have recommended initiating a biologic/subsequent entry biologic or switching to another biologic agent, and 3) who have internet access and email.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale | Change measure (baseline score compared to after using the ANSWER-2 intervention at month 1)
  The Decisional Conflict Scale (short version) measures personal perceptions of uncertainty in choosing options, factors contributing to uncertainty, and effective decision-making. It is one-dimensional and has 10 questions and three response categories (yes/no/unsure) used to compute one score.

SECONDARY OUTCOMES:
MeiQ | Change measure (baseline score compared to after using the ANSWER-2 intervention at month 1, and at month 2)
  The MeiQ consists of 6 subscales and a total of 29 items. MeiQ was developed and tested in three different samples of patients with rheumatic conditions on their knowledge of medications.
Partners in Health Scale | Change measure (baseline score compared to after using the ANSWER-2 intervention at month 1, and at month 2)
  The Partners in Health Scale is an 11-item measure, designed to assess self-efficacy, knowledge of RA and treatment, and self-management behaviours such as taking medication appropriately and adopting a healthy lifestyle.
Health Resource Utilization | Change measure (baseline score compared to after using the ANSWER-2 at month 2)
  The HRU questionnaire was developed for both self and interviewer administration in people with arthritis and other chronic conditions. It consists of a series of open-ended questions about individuals' visits to health professionals, use of investigative tests, hospital visits, use of medications, purchases of adaptive aids, and estimable productivity loss incurred by the individual and their caregivers due to the his/her health.

OTHER OUTCOMES:
CollaboRATE Scale | Change measure (baseline score compared to after using the ANSWER-2 intervention at month 1)
  a 3-item measure of the shared decision making process

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Professor
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of BC Study Website — http://arthritis.rehab.med.ubc.ca/2016/01/14/super-supporting-patient-care-with-electronic-resource/